CLINICAL TRIAL: NCT05180981
Title: Neuroimaging the Impact of Respiration and Respiratory-gated Neuromodulation on Human Glymphatic Physiology
Brief Title: Imaging Brain Fluids During Breathing
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Boston University Charles River Campus (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Laura Lewis, Assistant Professor, Boston University Charles River Campus
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 6029E; R01AT011429 (NIH)
Record Dates: First submitted 2021-11-03; First posted 2022-01-06 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Healthy
Keywords: Glymphatics; Cerebrospinal fluid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Breath task (Experimental): Participants will breathe in specific patterns.
  Interventions: Behavioral: Breathing task
- Transcutaneous vagal nerve stimulation (Experimental): Participants will receive transcutaneous vagal nerve stimulation in specific patterns.
  Interventions: Device: Transcutaneous vagal nerve stimulation; Behavioral: Breathing task

INTERVENTIONS:
Device: Transcutaneous vagal nerve stimulation — Noninvasive stimulation vs sham stimulation will be delivered via an auricular device.
  Arms: Transcutaneous vagal nerve stimulation
Behavioral: Breathing task — Participants will be asked to breathe in specific patterns.

SUMMARY:
This study will perform magnetic resonance imaging (MRI) measurements of hemodynamics and cerebrospinal fluid flow across breathing tasks and during breath-locked neuromodulation.

DETAILED DESCRIPTION:
Cerebrospinal fluid (CSF) flow is essential for brain health, as it clears waste products from the brain. This study will investigate how breathing affects the flow of CSF around the brain. The investigators will perform high resolution magnetic resonance imaging (MRI) scans in participants who are breathing in specific patterns or performing simple tasks and test the effects on CSF flow. Participants will complete an imaging study visit in which the investigators will image their brain activity while they perform simple tasks, including paced breathing tasks. The participants will be split into two arms: (1) paced breathing (25 participants low resolution, 15 participants high resolution), (2) transcutaneous vagal nerve stimulation (25 participants low resolution, 15 participants high resolution). The MRI scans will take place in the 7 Tesla MRI scanner at Massachusetts General Hospital.

ELIGIBILITY:
Inclusion Criteria:

* Adult age 18-70 years

Exclusion Criteria:

* No ferrous metal implanted in head or body
* No history of major head trauma
* No neurological or psychiatric disorder
* Not using medication that affects brain function
* No implanted electronic devices (e.g. pacemaker)
* No implant that poses an MR contraindication
* Not pregnant, suspect they are pregnant, or seeking to become pregnant
* Not claustrophobic
* No piercings or jewelry that cannot be removed
* Does not weigh more than 250 pounds
* Normal or contact-corrected normal vision

Exclusion for transcutaneous vagus nerve stimulation (tVNS) arm:

* Conditions of skin or anatomy that affect left auricle or forehead skin and could impact placement of electrodes for tVNS or forehead stimulation
* Diagnosis of significant cardiovascular or cerebrovascular disease [e.g. congestive heart failure, stroke, cardiac conduction disorders (including: bundle branch block, heart block, long Q-T syndrome), history of asystole or non-sustained ventricular tachycardia.
* Bradycardia (defined as resting heart rate <50 bpm)
* Hypotension defined as blood pressure <90/60 mmHg

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-01-18 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
functional magnetic resonance imaging (fMRI) signals | During study (2 hours)
  fMRI measures of hemodynamic responses. Units: percent signal change
Cerebrospinal fluid (CSF) signals | During study (2 hours)
  MR-based measures of CSF signals. Units: percent signal change

SECONDARY OUTCOMES:
Heart rate | During study ( 2 hours)
  Heart rate variability will be calculated. Units: milliseconds (ms)
Pulse oximetry | During study ( 2 hours)
  Amplitude of pulse oximetry signal. Units: arbitrary (no physical units are output by this system)
Respiratory physiology timing | During study (2 hours)
  Breath timing. Units: Hertz (Hz)
Respiratory physiology amplitude | During study (2 hours)
  Breath amplitude. Units: arbitrary (no physical units output by this sensor)

CONTACTS AND LOCATIONS:
Overall Officials: Laura Lewis, PhD, Principal Investigator — Boston University
Locations (2):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Boston University - Charles River Campus, Boston, Massachusetts